CLINICAL TRIAL: NCT06497114
Title: Validity and Reliability of the Egyptian-Arabic Version of ABILHAND-Kids in a Sample of Egyptian Children With Cerebral Palsy.
Brief Title: Validity and Reliability of the Egyptian-Arabic Version of ABILHAND-Kids
Status: Recruiting | Type: Observational
Sponsor: Horus University (Other)
Responsible Party: Principal Investigator, Amira Yosry El-Dwiny, lecturer of pediatric physical therapy, Horus University
Other Study IDs: P.T.REC/012/004994
Record Dates: First submitted 2024-07-04; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Cerebral Palsy
Keywords: hand function
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: ABILHAND-Kids questioner — questioner

SUMMARY:
HYPOTHESES It is hypothesized that the Egyptian-Arabic ABILHAND-Kids 21-item will be psychometrically appropriate to be used with Egyptian children with cerebral palsy.

DETAILED DESCRIPTION:
BACKGROUND Upper extremity functional impairment is a common problem in children with cerebral palsy. This has a significant impact on the children's manual ability which leads to activity limitation and participation restriction. The ABILHAND-Kids is a parent-reported outcome measure that quantifies the manual ability of children with CP. ABILHAND-Kids measures a child's ability to manage 21 daily activities that require the use of the upper limbs. The ABILHAND-Kids demonstrated very good measurement properties and is currently available in English, French, Dutch, Sweden, and Polish. It was also translated and adapted into the classic Arabic language in Saudi Arabia; in their study removal of two items resulted in a 19-item, valid, and reliable unidimensional scale meeting the requirement of the Rasch model without establishing measurement invariance between cultures. A linguistic adaptation is not sufficient to prove cross-cultural validity as item difficulties may vary across countries due to translation errors or cultural differences.

ELIGIBILITY:
Inclusion Criteria:

- Parents of 100 children with CP will be recruited.

Exclusion Criteria:

* mental retardation

Ages: 4 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: cerebral palsy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
ABILHAND-Kids | 4 months
  parent-reported outcome measure that quantifies the manual ability of children with CP.

CONTACTS AND LOCATIONS:
Locations (1):
- Horus University, Damietta, Egypt

IPD SHARING:
Plan to Share IPD: No